CLINICAL TRIAL: NCT01925794
Title: COBRA PZF™ Coronary Stent System in Native Coronary Arteries for Early Healing, Thrombus Inhibition, Endothelialization and Avoiding Long-Term Dual Anti-Platelet Therapy. The PzF Shield Trial
Brief Title: COBRA PZF™ Coronary Stent for Early Healing, Thrombus Inhibition, Endothelialization and Avoiding Long-Term DAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CeloNova BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COBRA 2012-01
Record Dates: First submitted 2013-08-09; First posted 2013-08-20 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
Keywords: Stent, Coronary Arteries for Early healing
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COBRA PzF Stent (Experimental): Single Arm study
  Interventions: Device: COBRA PzF

INTERVENTIONS:
Device: COBRA PzF

SUMMARY:
This is a prospective, multi-center, non-randomized, single arm clinical trial that will be conducted at up to 40 sites in the United States and Outside United States (OUS). This study will enroll patients with symptomatic ischemic heart disease due to a single de novo lesion contained within a native coronary artery with reference vessel diameter between 2.5 mm and 4.0 mm and lesion length ≤ 24 mm that is amenable to percutaneous coronary intervention (PCI) and stent deployment. All patients will be followed at 30 days, 6 months, 9 months, 1 year and annually for 5 years post index stenting procedure.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety and effectiveness of the COBRA PzF™ Coronary Stent System in the treatment of de novo lesions in native coronary arteries. The primary endpoint will be the incidence of target vessel failure (TVF, see definition below) within 270 days of treatment with the COBRA PzFTM Coronary Stent System. This rate will be compared to a performance goal derived using a meta-analysis from published historical data of the standard-of-care therapy, coronary stenting with bare metal stents.

PRIMARY STUDY HYPOTHESIS The CeloNova COBRA PzFTM Study will have a primary endpoint (TVF) rate less than 19.62% and by that will meet the performance goal for bare metal stents, per the results of the historical control group combined with relevant data for EXPRESS™, Driver™, Presillion/Presillion plus™ and NIRFLEX™ stents.

SECONDARY STUDY HYPOTHESIS The powered secondary endpoint for this trial is that the CeloNova COBRA PzFTM Study will have a 9-month in-stent late loss (LL) that meets or is lower than the performance goal of 1.1 mm.

NUMBER OF PATIENTS 296 patients will be enrolled to account for loss to follow-up, which is estimated to be approximately 5% (resulting in 281 evaluable patients), at up to 40 sites in United States and OUS. At least 40% of subjects will be enrolled in the United States.

PRIMARY ENDPOINT Target vessel failure (TVF), defined as cardiac death, target vessel myocardial infarction (MI) [Q wave or non-Q wave, ARC-definition], or clinically driven target vessel revascularization (TVR) by percutaneous or surgical methods within 270 days post-procedure.

SECONDARY ENDPOINTS

1. All Death at 30, 180, 270, 360, 720, 1080, 1440, and 1800 days
2. Cardiac Death at 30, 180, 270, 360, 720, 1080, 1440, and 1800 days
3. Major Adverse Cardiac Events (MACE), defined as cardiac death, MI (Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods at 30, 180, 270, 360, 720, 1080, 1440, and 1800 days
4. MI at 30, 180 and 270, 360, 720, 1080, 1440, and 1800 days CeloNova Biosciences, Inc. Confidential CeloNova COBRA PzF™ Study Protocol # COBRA 2012-01 6 07 May 14
5. Clinically driven TLR at 30, 180, 270, 360, 720, 1080, 1440, and 1800 days
6. Stroke (ischemic and hemorrhagic) at 30, 180, 270 and 360 days
7. Clinically driven TVR at 30, 180, 270 and 360 days
8. Composite Endpoint of Cardiac Death and MI at 30, 180, 270, and 360 days
9. TVF at 30, 180, and 360 days
10. Acute Success Rates

    1. Device Success: Attainment of < 30% final residual stenosis of the target lesion using only the COBRA PzFTM Coronary Stent System.
    2. Lesion Success: Attainment of < 30% final residual stenosis of the target lesion using any percutaneous method.
    3. Procedure Success: Attainment of < 30% final residual stenosis of the target lesion and no in-hospital MACE.
11. Bleeding or Vascular Complications at hospital discharge
12. Early Stent Thrombosis (ARC defined) at 30 days
13. Late Stent Thrombosis at 180, 270, and 360 days
14. Angiographic Endpoints (on first 90 evaluable patients) at 270 days (after clinical assessment)

    1. In-stent late loss (Secondary Endpoint hypothesis)
    2. In-segment percent diameter stenosis (%DS) (within the 5 mm margins proximal and distal to stent)
    3. In-stent percent diameter stenosis (%DS)
    4. In-segment late loss
    5. In-segment binary restenosis (stenosis of > 50% of the reference vessel diameter)
    6. In-stent binary restenosis
    7. In-stent minimum lumen diameter (MLD)
    8. In-segment MLD
    9. Longitudinal stent deformation
    10. Stent fracture
15. Optical Coherence Tomography Endpoints (on 45 subjects) at 270 days (after clinical assessment)

    1. in-stent neointimal thickness (NT)
    2. Lumen area
    3. Lumen volume
    4. Stent area
    5. Stent volume
    6. Proportion of uncovered and/or malopposed struts
    7. Stent fracture

ELIGIBILITY:
General Inclusion Criteria:

1. Patient >/= to 18 years old.
2. Eligible for percutaneous coronary intervention (PCI).
3. Patient understands the nature of the procedure and provides written informed consent prior to the catheterization procedure.
4. Patient is willing to comply with specified follow-up evaluation and can be contacted by telephone.
5. Acceptable candidate for coronary artery bypass graft (CABG) surgery.
6. Stable angina pectoris (Canadian Cardiovascular Society (CCS) 1, 2, 3 or 4) or unstable angina pectoris (Braunwald Class 1-3, B-C) or a positive functional ischemia study (e.g., ETT, SPECT, Stress echocardiography or Cardiac CT).
7. Male or non-pregnant female patient (Note: females of child bearing potential must have a negative pregnancy test prior to enrollment in the study).

Angiographic Inclusion Criteria

1. Patient indicated for elective stenting of a single stenotic lesion in a native coronary artery.
2. Reference vessel >/= 2.5 mm and </= 4.0 mm in diameter by visual estimate.
3. Target lesion </= 24 mm in length by visual estimate (the intention should be to cover the whole lesion with one stent of adequate length).
4. Protected left main lesion with >50% stenosis.
5. Target lesion stenosis >/= 70% and < 100% by visual estimate.
6. Target lesion stenosis <70% who meet physiological criteria for revascularization (i.e. positive FFR).

General Exclusion Criteria:

1. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
2. Previously enrolled in another stent trial within the prior 2 years.
3. ANY planned elective surgery or percutaneous intervention within the subsequent 3 months.
4. A previous coronary interventional procedure of any kind within 30 days prior to the procedure.
5. The patient requires staged procedure of either the target or any non-target vessel within 9 months post-procedure.
6. The target lesion requires treatment with a device other than PTCA prior to stent placement (such as, but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
7. Previous drug eluting stent (DES) deployment anywhere in the target vessel.
8. Any previous stent placement within 15 mm (proximal or distal) of the target lesion.
9. Co-morbid condition(s) that could limit the patient's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
10. Concurrent medical condition with a life expectancy of less than 12 months.
11. Documented left ventricular ejection fraction (LVEF) < 30% within 12 months prior to enrollment.
12. Patients with diagnosis of MI within 72 hours (i.e. CK-MB must be returned to normal prior to enrollment) or suspected acute MI at time of enrollment
13. Previous brachytherapy in the target vessel.
14. History of cerebrovascular accident or transient ischemic attack in the last 6 months.
15. Leukopenia (leukocytes < 3.5 x 10(9) / liter).
16. Neutropenia (Absolute Neutrophil Count < 1000/mm3) </= 3 days prior to enrollment.
17. Thrombocytopenia (platelets < 100,000/mm3) pre-procedure.
18. Active peptic ulcer or active GI bleeding.
19. History of bleeding diathesis or coagulopathy or inability to accept blood transfusions.
20. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, L-605 Cobalt chromium alloy or sensitivity to contrast media, which cannot be adequately pre-medicated.
21. Serum creatinine level > 2.0 mg/dl within 7 days prior to index procedure.
22. Patients unable to tolerate dual anti-platelets therapy (DAPT) for one month post procedure.

Angiographic Exclusion Criteria

1. Unprotected left main coronary artery disease (obstruction greater than 50% in the left main coronary artery that is not protected by at least one non-obstructed bypass graft to the LAD or Circumflex artery or a branch thereof).
2. Target vessel with any lesions with greater than 50% diameter stenosis outside of a range of 5 mm proximal and distal to the target lesion based on visual estimate or on-line QCA.
3. Target lesion (or vessel) exhibiting an intraluminal thrombus (occupying > 50% of the true lumen diameter) at any time.
4. Lesion location that is aorto-ostial or within 5 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX).
5. Target lesion with side branches > 2.0mm in diameter.
6. Target vessel is excessively tortuous (two bends > 90˚ to reach the target lesion).
7. Target lesion is severely calcified.
8. TIMI flow 0 or 1
9. Target lesion is in a bypass graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2013-08-21; Primary Completion 2015-11 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Cutlip, MD, Principal Investigator — Executive Director, Clinical Investigation, Harvard Clinical Research Institute; Sigmund Sliber, MD, Principal Investigator — Professor of Medicine at The University of Munich
Locations (35):
- United States (22):
  - Bakersfield Memorial Hospital, Bakersfield, California
  - Mt Sinai Medical Center, Miami Beach, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Heart Center of Indiana, Indianapolis, Indiana
  - Louisiana Heart Hospital, Lacombe, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - St Joseph's Hospital, Liverpool, New York
  - Lenox Hill Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Southern Oregon Cardiology, Medford, Oregon
  - York General Hospital, York, Pennsylvania
  - Cardiology Consultants of Texas, Dallas, Texas
  - Plaza Medical Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Cardiac Center, Lubbock, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - San Antonio Endovascular & Heart Institute, San Antonio, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Aspirus Heart & Vascular Institute, Wausau, Wisconsin
- France (6):
  - Clinique Axium, Aix-en-Provence
  - Hopital Henri Duffaut, Avignon
  - Albert Schweitzer Hospital, Colmar
  - Clinique du Diaconat, Mulhouse
  - Centre Hospitalier de Pau, Pau
  - Clinique St. Hilaire, Rouen
- Germany (2):
  - Sankt Kathatinen Hospital, Frankfurt
  - Kardiologische Praxis und Praxisklinik, München
- Paul Stradins Clinical University Hospital, Riga, Latvia
- Clinical Center of Serbia, Belgrade, Serbia
- Spain (2):
  - Hospital de la Santa Creu, Barcelona
  - Hospital Clinico San Carlos, Madrid
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was a total of 296 patients enrolled on this study between August 2013 - February 2015. A total of 35 clinical sites contributed the 296 patients enrolled.
Groups:
- COBRA PzF Stent: COBRA PzF Coronary Stent System
Period: 30 Days
Arm/Group | COBRA PzF Stent
Started | 296
Completed | 296
Not Completed | 0
Period: 180 Days
Arm/Group | COBRA PzF Stent
Started | 296
Completed | 292
Not Completed | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Period: 270 Days
Arm/Group | COBRA PzF Stent
Started | 292
Completed | 287
Not Completed | 5
Not completed — Death | 2
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.46 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 180
  Unknown or Not Reported | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan | 0
  Asian | 12
  Black or African American | 17
  Native Hawaiian or Pacific Islander | 0
  White or Caucasian | 206
  Other | 9
  Not reported | 52
Region of Enrollment [Count of Participants; unit: Participants]
  Latvia | 27
  United States | 166
  France | 44
  Serbia | 12
  Switzerland | 4
  Germany | 27
  Spain | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.46 (5.32)

OUTCOME MEASURES:

1. Primary Outcome: Target Vessel Failure (TVF)
Description: TVF defined as cardiac death, target vessel myocardial infarction (MI [Q wave or non-Q wave, ARC definition], or clinically driven target vessel revascularization (TVR) by percutaneous or surgical methods within 270 days post-procedure.
Time Frame: 270 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 290
percentage of participants | 11.38 [7.96 to 15.61]

2. Secondary Outcome: All Cause Mortality
Description: Death from any cause
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- COBRA PzF Stent: COBRA PzF Coronary Stent
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Participants | 1

3. Secondary Outcome: All Cause Mortality
Description: Death from any cause
Time Frame: 180 days
Population: The denominator is comprised of all the patients who had enough follow-up for 180-days analysis (at least 150 days allowing for 30 days window) or patients who had an event within 180 days post-procedure. The number of events varies for each of the endpoints resulting in different denominators.
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 294
Participants | 5

4. Secondary Outcome: All Cause Mortality
Description: Death from any cause
Time Frame: 270 days
Population: The denominator is comprised of all the patients who had enough follow-up for 270-days analysis (at least 240 days allowing for 30 days window) or patients who had an event within 270 days post-procedure. The number of events varies for each of the endpoints resulting in different denominators.
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 294
Participants | 6

5. Secondary Outcome: All Cause Mortality
Description: Death from any cause
Time Frame: 360 days
Population: The denominator is comprised of all the patients who had enough follow-up for 360-days analysis (at least 330 days allowing for 30 days window) or patients who had an event within 360 days post-procedure. The number of events varies for each of the endpoints resulting in different denominators.
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 291
Participants | 7

6. Secondary Outcome: All Cause Mortality
Description: Death from any cause
Time Frame: 1800 days
Population: The denominator is comprised of all the patients who had enough follow-up for 1800-days analysis (at least 1770 days allowing for 30 days window) or patients who had an event within 1800 days post-procedure. The number of events varies for each of the endpoints resulting in different denominators.
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 283
Participants | 34

7. Secondary Outcome: Cardiac Mortality
Description: Death due to any of the following:
  Acute myocardial infarction Cardiac perforation/pericardial tamponade Arrhythmia or conduction abnormality Cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure Death due to complication of a cardiac procedure including bleeding, vascular repair, transfusion reaction, or bypass surgery Any death is which a cardiac cause cannot be excluded
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Participants | 1

8. Secondary Outcome: Cardiac Mortality
Description: as for outcome 7
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 1

9. Secondary Outcome: Cardiac Mortality
Description: as for outcome 7
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 289
Participants | 1

10. Secondary Outcome: Cardiac Mortality
Description: as for outcome 7
Time Frame: 360 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 286
Participants | 1

11. Secondary Outcome: Cardiac Mortality
Description: as for outcome 7
Time Frame: 1800 days
Population: KM analysis estimate for patients in the ITT population who had enough follow-up for 1800-days analysis (at least 1770 days allowing for 30 days window) or patients who had an event within 1800 days post-procedure and censoring those not reaching the endpoint or sufficient follow up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 259
percentage of participants | 3.99 [1.68 to 6.29]

12. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: Cardiac death, MI (Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Participants | 19

13. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: as for outcome 12
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 23

14. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: as for outcome 12
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 289
Participants | 29

15. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: as for outcome 12
Time Frame: 360 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 286
Participants | 44

16. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: as for outcome 12
Time Frame: 1800 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 213
percentage of participants | 22 [17.2 to 26.8]

17. Secondary Outcome: Myocardial Infarction (MI-ARC Definition)
Description: Defined as either a Q wave MI (QWMI) or Non-Q wave MI (NQMI). QWMI is defined as development of new, pathological Q waves in 2 or more contiguous leads (as assessed by the Clinical Events Committee) with post-procedure CK-MB levels elevated above normal.
  NQWMI is defined as any elevation of post-procedure CK-MB to >=3 times site normal in the absence of pathological Q waves (historical definition). ARC definition includes Troponin or CK-MB >3 x UNL
Time Frame: 30 days
Population: The denominator is comprised of all the patients who had enough follow-up for 30-days analysis (at least 23 days allowing for 7 days window) or patients who had an event within 30 days post-procedure. The number of events varies for each of the endpoints resulting in different denominators.
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 295
Participants
  Q-wave MI | 0
  Non Q-wave MI | 18
  MI-ARC Definition | 18

18. Secondary Outcome: Myocardial Infarction (MI-ARC Definition)
Description: Defined as either a Q wave MI (QWMI) or Non-Q wave MI (NQMI). QWMI is defined as development of new, pathological Q waves in 2 or more contiguous leads (as assessed by the Clinical Events Committee) with post-procedure CK-MB levels elevated above normal.
  NQWMI is defined as any elevation of post-procedure CK-MB to >=3 times site normal in the absence of pathological Q waves
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 291
Participants
  Q-wave MI | 0
  Non Q-wave MI | 18
  MI-ARC Definition | 20

19. Secondary Outcome: Myocardial Infarction (MI-ARC Definition)
Description: as for outcome 18
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 288
Participants
  Q-wave MI | 0
  Non Q-wave MI | 18
  MI-ARC Definition | 20

20. Secondary Outcome: Myocardial Infarction (MI-ARC Definition)
Description: as for outcome 18
Time Frame: 360 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 285
Participants
  Q-wave MI | 0
  Non Q-wave MI | 21
  MI-ARC Definition | 24

21. Secondary Outcome: Myocardial Infarction (MI-ARC Definition)
Description: as for outcome 18
Time Frame: 1800 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 237
percentage of participants | 10.1 [6.62 to 13.6]

22. Secondary Outcome: Cardiac Death or MI (ARC Definition)
Description: Composite Endpoint of Cardiac Death or MI (ARC definition)
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Participants | 19

23. Secondary Outcome: Cardiac Death or MI (ARC Definition)
Description: Composite Endpoint of Cardiac Death and MI (ARC definition)
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 19

24. Secondary Outcome: Cardiac Death or MI (ARC Definition)
Description: Composite Endpoint of Cardiac Death or MI (ARC definition)
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 289
Participants | 19

25. Secondary Outcome: Cardiac Death or MI (ARC Definition)
Description: Composite Endpoint of Cardiac Death or MI (ARC definition)
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 286
Participants | 25

26. Secondary Outcome: Clinically Driven TLR
Description: Defined as a percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis of >= 50% by QCA, or revascularization of a target vessel with a diameter stenosis of >=70% by QCA without either angina or a positive functional study.
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 295
Participants | 0

27. Secondary Outcome: Clinically Driven TLR
Description: as for outcome 26
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 291
Participants | 7

28. Secondary Outcome: Clinically Driven TLR
Description: as for outcome 26
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 288
Participants | 13

29. Secondary Outcome: Clinically Driven TLR (Clinical and Angiographic Cohorts)
Description: as for outcome 26
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 285
Participants | 27

30. Secondary Outcome: Clinically Driven TLR (Clinical Cohorts)
Description: as for outcome 26
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 170
Participants | 8

31. Secondary Outcome: Clinically Driven TLR (Clinical and Angiographic Cohorts)
Description: as for outcome 26
Time Frame: 1800 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 228
percentage of participants | 12 [8.20 to 15.8]

32. Secondary Outcome: Clinically Driven TLR (Clinical Cohorts)
Description: as for outcome 26
Time Frame: 1800 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 139
percentage of participants | 7.76 [3.69 to 11.8]

33. Secondary Outcome: Clinically Driven TVR
Description: Defined as a percutaneous intervention or surgical bypass of any segment of the target vessel associated with positive functional ischemia study or ischemic symptoms AND an angiographic minimal lumen diameter stenosis >= 50% by QCA, or revascularization of a target vessel with diameter stenosis >=70% by QCA without either angina or a positive functional study.
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 295
Participants | 1

34. Secondary Outcome: Clinically Driven TVR
Description: as for outcome 33
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 291
Participants | 9

35. Secondary Outcome: Clinically Driven TVR
Description: as for outcome 33
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 289
Participants | 17

36. Secondary Outcome: Clinically Driven TVR
Description: as for outcome 33
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 286
Participants | 34

37. Secondary Outcome: Target Vessel Failure (TVF)
Description: TVF defined as cardiac death, target vessel myocardial infarction (MI) [Q wave or non-Q wave, ARC definition], or clinically driven target vessel revascularization (TVR) by percutaneous or surgical methods.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Participants | 20

38. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 37
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 25

39. Secondary Outcome: Target Vessel Failure (TVF)
Description: as for outcome 37
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 287
Participants | 50

40. Secondary Outcome: Stroke (Ischemic and Hemorrhagic)
Description: Defined as sudden onset of vertigo, numbness, dysphasia, weakness, visual field defects, dysarthria or other focal neurological deficits due to vascular lesions of the brain such as hemorrhage, embolism, thrombosis, or rupturing aneurysm, that persists more than 24 hours.
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 295
Participants | 0

41. Secondary Outcome: Stroke (Ischemic and Hemorrhagic)
Description: as for outcome 40
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 1

42. Secondary Outcome: Stroke (Ischemic and Hemorrhagic)
Description: as for outcome 40
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 289
Participants | 1

43. Secondary Outcome: Device Success
Description: Attainment of <30% final residual stenosis of the target lesion using only the COBRA PzF Coronary Stent System
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 291
Participants | 291

44. Secondary Outcome: Stroke (Ischemic and Hemorrhagic)
Description: as for outcome 40
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 286
Participants | 2

45. Secondary Outcome: Lesion Success
Description: Attainment of <30% final residual stenosis of the target lesion using any percutaneous method
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 254

46. Secondary Outcome: Procedure Success
Description: Attainment of <30% final residual stenosis of the target lesion and no in-hospital MACE
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 292
Participants | 241

47. Secondary Outcome: Bleeding or Vascular Complications
Description: Bleeding Complications: Procedure-related hemorrhagic event that requires a transfusion and/or surgical intervention Vascular Complications: May include pseudo aneurysm, arteriovenous fistula (AVF), peripheral ischemia/nerve injury, and vascular event requiring transfusion or surgical repair
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 296
Participants | 0

48. Secondary Outcome: Early Stent Thrombosis (ARC Definition)
Description: Early Stent Thrombosis (ARC Definition) 0-30 days post index procedure
Time Frame: 30 days
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 295
Participants | 0

49. Secondary Outcome: Late Stent Thrombosis
Description: Stent Thrombosis after 30 days and on or before 180 days
Time Frame: 180 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 291
Participants | 0

50. Secondary Outcome: Late Stent Thrombosis
Description: Stent Thrombosis after 30 days and on or before 270 days
Time Frame: 270 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 288
Participants | 0

51. Secondary Outcome: Late Stent Thrombosis
Description: Stent Thrombosis after 30 days and on or before 360 days
Time Frame: 360 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 285
Participants | 0

52. Secondary Outcome: Definite and Probable Stent Thrombosis
Description: as for outcome 26
Time Frame: 1800 days
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 259
percentage of participants | 0 [0 to 0]

53. Secondary Outcome: In-Segment Percent Diameter Stenosis
Description: Relative changes that occur in the percent diameter stenosis of the segment and are provided by the following relationship: % diameter stenosis= (1-[MLD/Reference diameter]) x 100
Time Frame: 270 days
Population: Angiographic subset included 115 of the 296 enrolled. Therefore, only 115 participants analyzed.
Measure: Mean (Standard Deviation); unit: percentage of vessel
Groups:
- Angiographic Cohort: A group of patients who underwent angiographic assessment after the clinical assessment at 270 days.
Arm/Group | Angiographic Cohort
Number analyzed (Participants) | 115
percentage of vessel
  In-Segment percent diameter stenosis (%DS) | 38.34 (17.03)
  In-Stent percent diameter stenosis (%DS) | 36.89 (18.30)

54. Secondary Outcome: In-Stent and In-Segment MLD and Late Loss
Description: * In-stent and in-Segment minimal lumen diameter obtained immediately after stent implantation and at angiographic assessment at 270 days.
  * In-stent or in-segment late loss was defined as the difference between minimum lumen diameter (in-stent or in-segment) immediately after implantation and that obtained at angiographic follow-up at 270 days.
Time Frame: 270 days
Population: Angiographic subset included 115 of the 296 enrolled. Therefore, the overall number of participants analyzed for this outcome measure is 115.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Angiographic Cohort: A group of patients who underwent an angiographic assessment after the clinical assessment at 270 days
Arm/Group | Angiographic Cohort
Number analyzed (Participants) | 115
mm
  In-Stent Late Loss | 0.83 (0.48)
  In-segment late loss | 0.52 (0.49)
  In-stent minimum lumen diameter | 1.78 (0.63)
  In-segment minimum lumen diameter | 1.72 (0.60)

55. Secondary Outcome: Angiographic Endpoints
Description: Angiographic subset included 115 of the 296 enrolled. Therefore, the overall number of participants analyzed for this outcome measure is 115.
Time Frame: 270 days
Population: Angiographic subset of patients
Measure: Number; unit: percentage of lesions
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 115
percentage of lesions
  In-segment binary restenosis | 28.57
  In-stent binary angiographic restenosis | 25.64
  Stent fracture | 0.00

56. Secondary Outcome: In-stent Neointimal Thickness (INT)
Description: in-stent neointimal thickness assessed by Optical Coherence Tomography
Time Frame: 270 days
Population: OCT subset included 57 of the 296 enrolled. Therefore, the overall number of participants analyzed for this outcome measure is 57.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- OCT Cohort: A group of those patients who underwent OCT assessment after the clinical follow up at 270 days
Arm/Group | OCT Cohort
Number analyzed (Participants) | 57
mm | 0.33 (0.15)

57. Secondary Outcome: Percentage of Uncovered and/or Malapposed Struts
Description: This measure assess the average proportion of uncovered and or malapposed struts measured by Optical Coherence Tomography in participants
Time Frame: 270 days
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: % of Uncovered and/or Malapposed Struts
Arm/Group | OCT Cohort
Number analyzed (Participants) | 57
% of Uncovered and/or Malapposed Struts | 0.00 (0.01)

58. Secondary Outcome: Lumen and Stent Area Measurements
Description: Optical Coherence Tomography assessment of the lumen and stent area after the clinical follow up at 270 days
Time Frame: 270 days
Population: OCT subset included only 57 of the 296 participants enrolled. Therefore, only 57 participants analyzed.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | OCT Cohort
Number analyzed (Participants) | 57
mm^2
  Lumen Area | 5.52 (2.52)
  Stent Area | 8.41 (2.69)

59. Secondary Outcome: Lumen and Stent Volume
Description: Optical Coherence Tomography assessment of the lumen and stent volume after the clinical follow up at 270 days
Time Frame: 270 days
Population: OCT subset includes 57 of the 296 enrolled. Therefore, only 57 participants analyzed.
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | COBRA PzF Stent
Number analyzed (Participants) | 57
mm3
  Lumen volume | 97.44 (61.27)
  Stent volume | 149.06 (75.99)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality assessed for 1800 days. Serious and Other Adverse Events assessed for 270 days
Arm/Group | COBRA PzF Stent
All-Cause Mortality (participants affected / at risk) | 34/283
Serious Adverse Events (participants affected / at risk) | 87/296
Other Adverse Events (participants affected / at risk) | 0/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COBRA PzF Stent (N=296)
Acute Coronary Syndrome (Cardiac disorders) | 4 (4)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 14 (15)
Angina Unstable (Cardiac disorders) | 1 (2)
Atrial Fibrillation (Cardiac disorders) | 8 (9)
Atrial Flutter (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 8 (9)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophagitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Impaired Healing (General disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 6 (7)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1)
Appendicitis Perforated (Infections and infestations) | 1 (1)
Necrotising Fasciitis (Infections and infestations) | 1 (1)
Nosocomial Infection (Infections and infestations) | 1 (1)
Oophoritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Salpingitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1)
Arterial Restenosis (Injury, poisoning and procedural complications) | 1 (1)
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 24 (25)
Post Pocedural Hematoma (Injury, poisoning and procedural complications) | 2 (2)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Blood Creatinine Phosphokinase Increased (Investigations) | 1 (1)
Cardiac Enzymes Increased (Investigations) | 1 (1)
Electrocardiogram Change (Investigations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Adenocarcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleural Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Parkinsonian Gait (Nervous system disorders) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Vascular Dementia (Nervous system disorders) | 1 (1)
Calculus Ureteric (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial Stenosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Intermittent Claudication (Vascular disorders) | 1 (2)
Peripheral Vascular Disorder (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less